CLINICAL TRIAL: NCT04296877
Title: Evaluation of Wear Experience With PRECISION1® Contact Lenses in Previous Acuvue® Oasys® Lens Wearers
Brief Title: Evaluation of Wear Experience With a Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jennifer Fogt, Associate Professor Clinical, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0019
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Contact Lens
Keywords: Daily Disposable Contact Lens; Soft Contact Lens; Spherical Contact Lens

STUDY DESIGN:
Intervention Model Description: This is a single arm, non-comparative study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All study participants (Experimental): All subjects are fit into daily disposable contact lenses after wearing their optimized habitual contact lenses for ~ 1 week. Subjects are requested to wear the lenses for two weeks, for a minimum of at least 6 hours per day for 10 days.
  Interventions: Device: Daily Disposable Contact Lens

INTERVENTIONS:
Device: Daily Disposable Contact Lens — Soft, daily disposable spherical contact lens used to correct distance vision.

SUMMARY:
To evaluate the wear experience of current two-week contact lens wearers after they have been fit into a daily disposable contact lens. This is a single arm, non-comparative study.

DETAILED DESCRIPTION:
This is a single arm, non-comparative study. All participants were habitual lens wearers of the same brand of lenses, and were re-fit with the study lenses.

ELIGIBILITY:
Inclusion Criteria:

* Must be current Acuvue® Oasys® spherical contact lens wearers.
* Distance visual acuity of 20/25 or better with current contact lenses.
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI).
* Ability to give informed consent.
* Willing to spend time for the study, which includes attending two study visits and wearing contact lenses on days between study visits.
* Either gender.
* Any racial or ethnic origin.

Exclusion Criteria:

* No current ocular inflammation or infection.
* Not currently pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fogt, OD, MS, Principal Investigator — The Ohio State University College of Optometry
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Study: All subjects are re-fit into their habitual reusable soft contact lenses to optimize vision. Subjects are requested to wear the lenses for one week, for a minimum of at least 6 hours per day for 5 days.
  Subjects then return and are fit with the daily disposable soft contact lens. After wearing the daily disposable lenses, participants return to assess vision and lens fit and answer surveys about their experience.
Period: Overall Study
Arm/Group | Single Arm Study
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants
Groups:
- All Participants Wear Study Daily Disposable Contact Lenses: All subjects are re-fit into their habitual reusable soft contact lenses to optimize vision. Subjects are requested to wear the lenses for one week, for a minimum of at least 6 hours per day for 5 days.
  Subjects then return and are fit with the daily disposable soft contact lens. After wearing the daily disposable lenses, participants return to assess vision and lens fit and answer surveys about their experience.
Arm/Group | All Participants Wear Study Daily Disposable Contact Lenses
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens Dry Eye Questionnaire (CLDEQ-8) Survey
Description: Participants complete the Contact Lens Dry Eye Questionnaire (CLDEQ-8) survey. This is an 8 question survey assesses symptoms while wearing contact lenses with possible scores from 0 (no symptoms) to 37 (maximum symptoms). Higher scores indicate worsening symptoms of dry eye while wearing lenses.
Time Frame: 2 weeks
Population: All subjects were in the same arm, and wore both types of lenses. This was not a comparative study.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- All Study Participants: All subjects are re-fit into their habitual reusable soft contact lenses to optimize vision. Subjects are requested to wear the lenses for one week, for a minimum of at least 6 hours per day for 5 days.
  Subjects then return and are fit with the daily disposable soft contact lens. After wearing the daily disposable lenses, participants return to assess vision and lens fit and answer surveys about their experience.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
units on a scale | 9.5 [6 to 17.75]

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- All Study Participants: All subjects are re-fit into their habitual reusable soft contact lenses to optimize vision. Subjects are requested to wear the lenses for one week, for a minimum of at least 6 hours per day for 5 days.
  Subjects then return and are fit with the daily disposable soft contact lens. After wearing the daily disposable lenses, participants return to assess vision and lens fit and answer surveys about their experience.
  Adverse events were not collected separately for the habitual reusable lenses and daily disposable lenses.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT04296877/Prot_SAP_000.pdf